CLINICAL TRIAL: NCT04987606
Title: POST COvid-19 Interstitial Lung DiseasE (POSTCODE) A Study of Genetic and Environmental Interactions: an Observational Cohort Study.
Brief Title: Post COVID-19 Interstitial Lung Disease: A Study of Genetic and Environmental Interactions
Acronym: POSTCODE
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 21SM6765
Record Dates: First submitted 2021-07-19; First posted 2021-08-03 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Pulmonary Fibrosis; COVID-19 Pneumonia
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to understand why some people who have had COVID-19 develop scarring of the lungs and why some people recover more quickly than others.

DETAILED DESCRIPTION:
A large number of people diagnosed with COVID-19 suffer from long term symptoms, predominantly breathlessness and fatigue whether or not they were admitted to hospital. While there are a number of causes of long-term breathlessness following COVID-19 one of the most common, and potentially concerning with regards to long term prognosis is Interstitial Lung Disease.

The fibrogenic potential of SARS-CoV-2 is currently unknown but is predicted to be substantial based on the experience of previous coronavirus outbreaks and emerging data from this pandemic.

The investigators do not yet understand how scarring occurs following SARS-CoV-2, nor why there is resolution in some individuals and persistent or progressive disease in others. The investigators therefore plan to undertake bronchoscopy (camera test into the lungs) to examine for changes in the way the cells lining the lung behave, using genetics, and differences in the bacteria living in the airways in patients whom have developed scarring following COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of SARS-CoV-2 PCR/Seropositive
* Presence of interstitial lung disease on CT
* Participant is willing and able to give informed consent for participation in the study
* Aged 18 years or above

Exclusion Criteria:

* Confirmed ILD diagnosis prior to March 2020
* Patients with co-morbid disease that in the opinion of the investigators gives them an expected life expectancy of less than one year will be excluded from the study.
* Use of steroids at baseline visit

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with interstitial lung disease following COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Differences in the bacterial burden and composition of the respiratory microbiome in post covid fibrosis compared to health | 2 years
  The lower airway bacterial burden and microbiome will be characterised in patients with post covid fibrosis and compared to that of health.

SECONDARY OUTCOMES:
Change in bacterial burden over time in post covid fibrosis | 2 years
  Differences in the airway bacterial burden at baseline and one year following covid-19 infection

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - University College London NHS Foundation Trust, London
  - Royal Brompton Hospital, London
  - Imperial College Healthcare Trust, London
  - Manchester University NHS Trust, Manchester